CLINICAL TRIAL: NCT01235754
Title: A Phase III, Multi-Center Extension Study to Assess Persistence of Benefit of LibiGel for the Treatment of Hypoactive Sexual Desire Disorder (HSDD) in Surgically Menopausal Women
Brief Title: Extension Study to Assess Persistence of Benefit of LibiGel for the Treatment of Hypoactive Sexual Desire Disorder (HSDD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioSante Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TESTW009
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Hypoactive Sexual Desire Disorder
Keywords: testosterone; hypoactive sexual desire disorder; menopause
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo gel (Placebo Comparator): placebo transdermal gel
  Interventions: Drug: placebo gel
- testosterone gel (Experimental): transdermal testosterone gel
  Interventions: Drug: transdermal testosterone gel 1%

INTERVENTIONS:
Drug: transdermal testosterone gel 1% — 300 mcg once daily transdermal testosterone gel 1%
  Other Names: LibiGel transdermal testosterone gel 1%
  Arms: testosterone gel
Drug: placebo gel — once daily transdermal placebo gel
  Other Names: transdermal placebo gel
  Arms: placebo gel

SUMMARY:
The objective of this study is to evaluate the persistence of benefit of LibiGel (testosterone gel) 300 mcg/day compared to placebo gel in a 12 week post-treatment period of Hypoactive Sexual Desire Disorder (HSDD) in surgically menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* must have completed a minimum of 22 weeks of the 24-week TESTW006 or TESTW008 clinical trial

Exclusion Criteria:

* Any condition (including a change in sexual or relationship history) that would make the subject unsuitable for participation in the trial in the opinion of the Investigator

Ages: 30 Years to 66 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in the 4-week total number of days with at least one satisfying sexual event from the baseline period (during the previous study) to weeks 9-12 of the current study | 12 weeks
  This study is to assess the persistence of benefit following the withdrawal of testosterone gel (LibiGel) in the treatment of Hypoactive Sexual Desire Disorder (HSDD) in healthy, surgically menopausal women.

SECONDARY OUTCOMES:
change from baseline (previous study) in the mean FSDS-R question 13 score to week 12 of the current study | 12 weeks
  This study is to acess the persistence of benefit following the withdrawal of testosterone gel 1% (LibiGel)in the treatment of Hypoactive Sexual Desire Disorder (HSDD) in healthy, surgically menopausal women.
change from baseline (previous study) in the total number of days with at least one satisfying sexual event at weeks 4 and 8 of the current study | 12 weeks
  This study is to assess the persistence of benefit following the withdrawal of testosterone gel (LibiGel)in the treatment of Hypoactive Sexual Desire Disorder (HSDD) in healthy, surgically menopausal women.

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Snabes, MD, PhD, Study Director — BioSante Pharmaceuticals
Locations (102):
- United States (98):
  - BioSante Site #095, Hoover, Alabama
  - BioSante Site #014, Huntsville, Alabama
  - BioSante Site #146, Mobile, Alabama
  - BioSante Site #171, Chandler, Arizona
  - BioSante Site #145, Glendale, Arizona
  - BioSante Site #027, Glendale, Arizona
  - BioSante Site #121, Phoenix, Arizona
  - BioSante Site #137, Tucson, Arizona
  - BioSante Site #052, Hot Springs, Arkansas
  - BioSante Site #155, Little Rock, Arkansas
  - BioSante Site #221, Berkeley, California
  - BioSante Site #182, Buena Park, California
  - BioSante Site #162, Sacramento, California
  - BioSante Site #008, San Diego, California
  - BioSante Site #159, Walnut Creek, California
  - BioSante Site #007, Denver, Colorado
  - BioSante Site #026, Lakewood, Colorado
  - BioSante Site #132, New Britain, Connecticut
  - BioSante Site #151, New London, Connecticut
  - BioSante Site #036, Ridgefield, Connecticut
  - BioSante Site #143, Jacksonville, Florida
  - BioSante Site #024, Miami, Florida
  - BioSante Site #111, Orlando, Florida
  - BioSante Site #219, Pinellas Park, Florida
  - BioSante Site #041, St. Petersburg, Florida
  - BioSante Site #009, West Palm Beach, Florida
  - BioSante Site #115, Atlanta, Georgia
  - BioSante Site #141, Roswell, Georgia
  - BioSante Site #202, Idaho Falls, Idaho
  - BioSante Site #017, Meridian, Idaho
  - BioSante Site #189, Addison, Illinois
  - BioSante Site #133, Chicago, Illinois
  - BioSante Site #167, Newburgh, Indiana
  - BioSante Site #163, Overland Park, Kansas
  - BioSante Site #214, Lexington, Kentucky
  - BioSante Site #110, Metarie, Louisiana
  - BioSante Site #005, Shreveport, Louisiana
  - BioSante Site #206, Fall River, Massachusetts
  - BioSante Site #035, Ann Arbor, Michigan
  - BioSante Site #124, Bingham Farms, Michigan
  - BioSante Site #044, Detroit, Michigan
  - BioSante Site #047, Grand Rapids, Michigan
  - BioSante Site #105, Kalamazoo, Michigan
  - BioSante Site #033, Saginaw, Michigan
  - BioSante Site #031, Saint Clair Shores, Michigan
  - BioSante Site #208, Edina, Minnesota
  - BioSante Site #198, Saint Paul, Minnesota
  - BioSante Site #104, St Louis, Missouri
  - BioSante Site #127, Billings, Montana
  - BioSante Site #051, Missoula, Montana
  - BioSante Site #006, Lincoln, Nebraska
  - BioSante Site #015, Poughkeepsie, New York
  - BioSante Site #059, Cary, North Carolina
  - BioSante Site #107, Raleigh, North Carolina
  - BioSante Site #131, Winston-Salem, North Carolina
  - BioSante Site #056, Fargo, North Dakota
  - BioSante Site #210, Akron, Ohio
  - BioSante Site #130, Beachwood, Ohio
  - BioSante Site #212, Cincinnati, Ohio
  - BioSante Site #101, Cleveland, Ohio
  - BioSante Site #213, Columbus, Ohio
  - BioSante Site #160, Englewood, Ohio
  - BioSante Site #153, Gallipolis, Ohio
  - BioSante Site #138, West Chester, Ohio
  - BioSante Site #129, Tulsa, Oklahoma
  - BioSante Site #050, Eugene, Oregon
  - BioSante Site #106, Eugene, Oregon
  - BioSante Site #126, Medford, Oregon
  - BioSante Site #165, Jenkintown, Pennsylvania
  - BioSante Site #099, Sellersville, Pennsylvania
  - BioSante Site #197, Wexford, Pennsylvania
  - BioSante Site #117, Anderson, South Carolina
  - BioSante Site #089, Columbia, South Carolina
  - BioSante Site #209, Greer, South Carolina
  - BioSante Site #049, Watertown, South Dakota
  - BioSante Site #069, Chattanooga, Tennessee
  - BioSante Site #078, Memphis, Tennessee
  - BioSante Site #042, Nashville, Tennessee
  - BioSante Site #120, North Jackson, Tennessee
  - BioSante Site #048, Austin, Texas
  - BioSante Site #073, Corpus Christi, Texas
  - BioSante Site #220, Dallas, Texas
  - BioSante Site #147, Dallas, Texas
  - BioSante Site #039, Houston, Texas
  - BioSante Site #122, Houston, Texas
  - BioSante Site #154, Hurst, Texas
  - BioSante Site #211, San Antonio, Texas
  - BioSante Site #218, Murray, Utah
  - BioSante Site #144, Pleasant Grove, Utah
  - BioSante Site #102, Salt Lake City, Utah
  - BioSante Site #096, Williston, Vermont
  - BioSante Site #003, Charlottesville, Virginia
  - BioSante Site #086, Norfolk, Virginia
  - BioSante Site #053, Richmond, Virginia
  - BioSante Site #083, Mountlake Terrace, Washington
  - BioSante Site #128, Seattle, Washington
  - BioSante Site #181, Tacoma, Washington
  - BioSante Site #183, Walla Walla, Washington
- Canada (4):
  - BioSante Site# 123, Ottawa, Ontario
  - BioSante Site #188, Sarnia, Ontario
  - BioSante Site #054, Windsor, Ontario
  - BioSante Site #193, Shawinigan, Quebec